CLINICAL TRIAL: NCT05112939
Title: A Phase 1, Single-blind, Randomized, Parallel-group Study in Healthy Participants to Investigate the Single-dose Pharmacokinetics, Safety and Tolerability of Rilpivirine After Subcutaneous Administration of a Rilpivirine Extended-Release Suspension Alone, and of Rilpivirine and Cabotegravir After Co-administration With Cabotegravir Extended-Release Suspension
Brief Title: A Study of a Rilpivirine Extended-Release Suspension in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR109089; TMC278LAHTX1003 (Other: Janssen Research & Development, LLC); 2021-002697-31 (EudraCT Number)
Expanded Access: NCT03847376 (Approved for marketing)
Record Dates: First submitted 2021-11-02; First posted 2021-11-09 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Healthy
MeSH Terms: interventions — Rilpivirine; cabotegravir

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Panel A: Rilpivirine (RPV) Long-acting (LA) (Experimental): Participants will receive one dose of RPV LA (formulation 1) under different conditions (Treatment A and B) on Day 1.
  Interventions: Drug: RPV LA
- Panel B: RPV LA (Experimental): Participants will receive one dose of RPV LA (formulation 2) under different conditions (Treatment C and D) on Day 1.
  Interventions: Drug: RPV LA
- Panel C: RPV LA (Experimental): Participants will receive one dose of RPV LA (formulation 1) under different conditions (Treatment E and F) on Day 1, based on interim data of Panel A.
  Interventions: Drug: RPV LA
- Panel D: RPV LA (Experimental): Participants will receive one dose of RPV LA (formulation 2) under different conditions (Treatment G and H) on Day 1, based on interim data of Panel B.
  Interventions: Drug: RPV LA
- Panel E: RPV LA + Cabotegravir (CAB) LA (Experimental): Participants will receive one dose of RPV LA (formulation 1) with CAB LA (formulation 3) (Treatment I) on Day 1.
  Interventions: Drug: RPV LA; Drug: CAB LA

INTERVENTIONS:
Drug: RPV LA — RPV LA will be administered at different formulations.
  Other Names: TMC278
Drug: CAB LA — CAB LA will be administered at formulation 3.
  Other Names: GSK1265744
  Arms: Panel E: RPV LA + Cabotegravir (CAB) LA

SUMMARY:
The purpose of this study is to characterize the single dose pharmacokinetics (PK) and evaluate the safety and tolerability of subcutaneous administration of rilpivirine (RPV) long-acting (LA) or RPV LA in combination with cabotegravir (CAB) LA extended release suspensions in different conditions in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) (based on the average value of triplicate ECGs) performed at screening (results must be available on Day -1)
* Participant must be healthy on the basis of clinical laboratory tests performed at screening (results must be available prior to dosing on Day 1). If there are abnormalities, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the investigator
* All women participants must have a negative highly sensitive serum (Beta-human chorionic gonadotropin [Beta-hCG]) pregnancy test at screening and on Day -1
* A woman must agree not to donate eggs (ova, oocytes) or freeze for future use for the purposes of assisted reproduction during the study and for at least 72 weeks after receiving the dose of study intervention
* A male participant (not vasectomized) who is heterosexually active with a woman of childbearing potential must agree to use two effective contraceptive methods for the duration of the study (72 weeks follow-up), or for at least 72 weeks after receiving the dose of study intervention for those who do not complete the study

Exclusion Criteria:

* Participant with a history of or current illness that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study intervention to the participant or that could prevent, limit or confound the protocol specified assessments. This may include, but is not limited to, hepatic or renal dysfunction, cardiac disease, vascular, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, neurologic, hematologic, coagulation disorders (including any abnormal bleeding or blood dyscrasias), or psychiatric disturbances
* Participant has a history of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, which is considered cured with minimal risk of recurrence)
* Participant has known allergies, hypersensitivity, or intolerance to Cabotegravir (CAB) or its excipients
* Participants with the following ECG findings, if clinically significant: abnormal PR, QRS, and QTc intervals; rhythm abnormalities; evidence of acute ischemic changes
* Participants with a history of clinically relevant skin disease such as, but not limited to, dermatitis, eczema, drug rash, drug allergy, psoriasis, food allergy, urticaria

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Plasma Concentration of Rilpivirine (RPV) | Up to 72 weeks
  Plasma samples will be analyzed to determine concentrations of RPV using a validated, specific, and sensitive method.
Plasma Concentration of Cabotegravir (CAB) | Up to 72 weeks
  Plasma samples will be analyzed to determine concentrations of CAB using a validated, specific, and sensitive method.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Up to 72 weeks
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/ biological agent under study.
Number of Participants with Injection-Site Reactions | Up to 72 weeks
  Number of participants with injection-site reactions will be reported. A study intervention injection-site reaction is any adverse reaction at a subcutaneous study intervention injection-site.
Number of Participants with Abnormalities in 12-Lead Electrocardiograms (ECGs) | Up to 72 weeks
  Number of participants with abnormalities in 12- lead ECGs (heart rate, PR, QRS and QT corrected [QTc]) will be reported.
Pain Assessment using Visual Analogue Scale (VAS) | Up to 72 weeks
  Pain assessments will be performed by collecting pain intensity scores using 100-millimetre (mm) VAS.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (3):
- United States (2):
  - PRA Health Sciences, Lenexa, Kansas
  - PRA Health Sciences, Salt Lake City, Utah
- PRA Health Sciences, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency